CLINICAL TRIAL: NCT05371353
Title: Evaluating the Immune Persistence of Recombination Quadrivalent HPV Vaccine (Type 6, 11, 16, 18) in Healthy Chinese Female Subjects Aged 9 to 45 Years: A Phase 3, Open-label, Non-randomized Clinical Trial
Brief Title: Immune Persistence After the Whole Vaccination Shcedule With Recombination Quadrivalent HPV Vaccine
Status: Recruiting | Type: Observational
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 4-HPV-3003
Record Dates: First submitted 2022-05-04; First posted 2022-05-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: HPV Infections; Cervical Cancer Stage IIa; Vaginal Cancer; Genital Wart; CIN1; CIN2; CIN3
Keywords: Human papillomavirus; vaccine; Cervical Cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Vaginal Neoplasms; Condylomata Acuminata

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To access the immune persistence of Chinese women aged 9-45 years after receiving quadrivalent HPV vaccine with the immunization schedule of 0, 2 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in the phase III clinical trial of non inferior efficacy of HPV tetravalent vaccine of Yangchun Center for Disease Control and Prevention (protocol No.: 4-HPV-3001), completed three doses of HPV quadrivalent vaccine and provided blood sample at months 7; Or subjects who have participated in the bridging study of HPV quadrivalent vaccine of Mianyang Center for Disease Control and Prevention (scheme No.: 4-HPV-3002), completed the whole vaccine schedule at month 0，2，6, and provided blood sample at months 7;
* The subjects aged 9 to 17 years old at Mianyang site and their legal guardian should provide legal indentification; the subjects aged over 18 years old should provide legal indentification;
* The subject voluntarily agrees to enroll in this study. If the subject is a minor, both the subject and subject's legal guardian should voluntarily agree to enroll in this study and sign an informed consent form;
* Be able to understand the study procedures and promise to participate in regular follow-ups under the requirements.

Exclusion Criteria:

* Enrolling or plan to enroll in other clinical trials (drugs or vaccines) (except that the observational clinical study and the subjects at Mianyang site are still in the post exemption safety follow-up stage of the 4-HPV-3002 trial);
* Suffering from thrombocytopenia or any coagulation dysfunction that can be a contraindication to blood collection (such as coagulation factor deficiency, coagulation diseases, platelet abnormalities, etc.);
* According to the investigator's judgment, the subject has any condition may interfere with process of evaluation of immune persistence.

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects aged 9-45 years old have completed receiving three doses of quadrivalent HPV vaccine and provided blood sample at month 7
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-05-14 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate (SCR) for Each of the HPV Types Contained in the Vaccine | Month 12
  The primary immue persistence outcome to evaluate respinses quadrivalent HPV vaccine was Year 5 seroconversion rate against HPV-types 6,11,16, and 18
SCR for Each of the HPV Types Contained in the Vaccine | Month 24
  The primary immue persistence outcome to evaluate respinses quadrivalent HPV vaccine was Year 5 seroconversion rate against HPV-types 6,11,16, and 18
SCR for Each of the HPV Types Contained in the Vaccine | Month 36
  The primary immue persistence outcome to evaluate respinses quadrivalent HPV vaccine was Year 5 seroconversion rate against HPV-types 6,11,16, and 18
SCR for Each of the HPV Types Contained in the Vaccine | Month 48
  The primary immue persistence outcome to evaluate respinses quadrivalent HPV vaccine was Year 5 seroconversion rate against HPV-types 6,11,16, and 18
SCR for Each of the HPV Types Contained in the Vaccine | Month 60
  The primary immue persistence outcome to evaluate respinses quadrivalent HPV vaccine was Year 5 seroconversion rate against HPV-types 6,11,16, and 18
Geometric Mean Titers (GMTs) for Each of the HPV Types Contained in the Vaccine | Month 12
  The primary immune persistence endpoint is anti-HPV type 6,11,16,and 18 antibody GMTs 5 years post dose 1 assessed among the subjects who were seropositive at Month 7
GMTs for Each of the HPV Types Contained in the Vaccine | Month 24
  The primary immune persistence endpoint is anti-HPV type 6,11,16,and 18 antibody GMTs 5 years post dose 1 assessed among the subjects who were seropositive at Month 7
GMTs for Each of the HPV Types Contained in the Vaccine | Month 36
  The primary immune persistence endpoint is anti-HPV type 6,11,16,and 18 antibody GMTs 5 years post dose 1 assessed among the subjects who were seropositive at Month 7
GMTs for Each of the HPV Types Contained in the Vaccine | Month 48
  The primary immune persistence endpoint is anti-HPV type 6,11,16,and 18 antibody GMTs 5 years post dose 1 assessed among the subjects who were seropositive at Month 7
GMTs for Each of the HPV Types Contained in the Vaccine | Month 60
  The primary immune persistence endpoint is anti-HPV type 6,11,16,and 18 antibody GMTs 5 years post dose 1 assessed among the subjects who were seropositive at Month 7

CONTACTS AND LOCATIONS:
Overall Officials: Jikai Zhang, Study Director — Guangdong Center for Disease Prevention and Control
Locations (2):
- China (2):
  - Yangchun Center For Disease Prevention And Control, Yangchun, Guangdong
  - Center for Disease Control and Prevention, Mianyang, Sichuan